CLINICAL TRIAL: NCT03329469
Title: The Value of Fractional Flow Reserve Derived From Coronary CT Angiography as Compared to CCTA or CCTA and Stress MPI in the Triage of Low to Intermediate Emergent Chest Pain Patients With Toshiba CT-FFR
Brief Title: The Value of CT-FFR Compared to CCTA or CCTA and Stress MPI in Low to Intermediate Risk ED Patients With Toshiba CT-FFR
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Northwell Health (Other)
Collaborators: Toshiba America Medical Systems, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Poon, Chief, Non-invasive Cardiac Imaging;System Director of Research, Cardiac Imaging, and Clinical Transformation, Northwell Health
Other Study IDs: Northwell IRB #17-0187
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease; Chest Pain; Acute Coronary Syndrome; Acute Myocardial Infarction
Keywords: Computed Tomography Fractional Flow Reserve (CT-FFR),; Computed Coronary Tomography Angiography (CCTA); Invasive Fractional Flow Reserve (iFFR); Fractional Flow Reserve (FFR); Emergency Department (ED); Emergency Room (ER)
MeSH Terms: conditions — Coronary Artery Disease; Chest Pain; Acute Coronary Syndrome; Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Experimental: 1: Toshiba CT-FFR Arm: All patients who consent will receive Toshiba CT-FFR and medically acceptable care based on the study protocol, commonly accepted standards of care, and the patients condition.
  Interventions: Device: Toshiba CT-FFR

INTERVENTIONS:
Device: Toshiba CT-FFR — Patients receiving CCTA to diagnose acute chest pain or unstable angina will receive CT-FFR to estimate rate of blood flow through the coronary arteries. The rate of flow will be compared to the rate found on Invasive FFR (the gold standard) if the subject receives invasive FFR.
  Other Names: Noninvasive CT-FFR, FFR-CT, Noninvasive FFR-CT

SUMMARY:
Coronary Computed Tomography Angiogram (CCTA) is a non-invasive imaging modality that has high sensitivity and negative predictive value for the detection of coronary artery disease (CAD). The main limitations of CCTA are its poor specificity and positive predictive value, as well as its inherent lack of physiologically relevant data on hemodynamic significance of coronary stenosis, a data that is provided either by non-invasive stress tests such as myocardial perfusion imaging (MPI) or invasively by measurement of the Fractional Flow Reserve (FFR). Recent advances in computational fluid dynamic techniques applied to standard CCTA are now emerging as powerful tools for virtual measurement of FFR from CCTA imaging (CT-FFR). These techniques correlate well with invasively measured FFR [1-4]. The primary purpose of this study is to evaluate the incremental benefit CT-FFR as compared to CCTA in triaging chest pain patients in emergency settings who are found to have obstructive CAD upon CCTA (generally >= 30% stenosis). Invasive FFR and short term clinical outcomes (90 days) will be correlated with each diagnostic modality in order to evaluate positive and negative predictive value of each.

Patients will undergo a CCTA, as part of routine emergency care. If the patient consents to participate in the study, the CCTA study will be assessed by Toshiba Software, to provide a computerized FFR reading, based on the CCTA study. If the noninvasive FFR diagnosis indicates obstructive disease, the patient will undergo cardiac catheterization with invasive FFR.

As CCTA utilization increases, the need to train additional imaging specialists will increase. This study will assess the capability of FFR-CT to enhance performance on both negative and positive predictive value for less experienced readers by providing feedback based on CT-FFR evaluation. If the use of CT-FFR improves accuracy of CCTA, as compared to the gold standard, (Invasive FFR), use of CT-FFR can potentially enhance performance for less experienced readers.

DETAILED DESCRIPTION:
Background:

Coronary Computed Tomography Angiogram (CCTA) is a non-invasive imaging modality that has high sensitivity and negative predictive value for the detection of coronary artery disease (CAD). The main limitations of CCTA are its poor specificity and positive predictive value, as well as its inherent lack of physiologically relevant data on hemodynamic significance of coronary stenosis, a data that is provided either by non-invasive stress tests such as myocardial perfusion imaging (MPI) or invasively by measurement of the Fractional Flow Reserve (FFR). Recent advances in computational fluid dynamic techniques applied to standard CCTA are now emerging as powerful tools for virtual measurement of FFR from CCTA imaging (CT-FFR). These techniques correlate well with invasively measured FFR [1-4]. The primary purpose of this study is to evaluate the incremental benefit CT-FFR as compared to CCTA in triaging chest pain patients in ED settings who are found to have obstructive CAD upon CCTA (generally > 30% and < 90% stenosis). Invasive FFR and short term clinical outcomes (90 days) will be correlated with each diagnostic modality in order to evaluate positive and negative predictive value of each when used incrementally with CCTA.

Investigational Agent:

CCTA is increasingly becoming a preferred non-invasive imaging modality because of its high sensitivity and negative predictive value for the detection of CAD. It has been shown to be a robust imaging modality for evaluation of chest pain, and is associated with decreased unnecessary hospital admission, length of stay, major adverse cardiovascular event rates, recidivism rates, and downstream resource utilization compared to standard evaluation [5]. While findings so far are highly suggestive of CCTA's significance as a gatekeeper for ICA by ruling out obstructive CAD, fewer than half of obstructive stenosis identified by CCTA are ischemia-causing, signifying its poor positive predictive value and inherent lack of physiological information [6-8]. Consequently, utilization of CCTA has not entirely averted need for downstream testing for functional assessment of CCTA-detected obstructive lesions either by stress testing or ICA. Recently a major treatment modality, associated with the use of CCTA, has become available that offers promise for improving positive predictive value and physiological relevant hemodynamic data. Advances in computational fluid dynamic techniques applied to standard CCTA are now emerging as a powerful tool for virtual measurement of FFR from CCTA imaging (CT-FFR). This technique correlates well with invasively measured FFR [1-4]. While HeartFlow, Inc. has established an FDA approved process to assess coronary artery flow using noninvasive CT-FFR, this data requires 24 to 48 hours for processing.

Toshiba CT-FFR processing is non-FDA approved. The analytic method for vessel evaluation differs from that used by HeartFlow. Currently Toshiba is operating studies at four organizations around the world to assess the product's performance. Recently, the company published results from a study conducted Australia that showed positive findings on a sample of 42 patients, with positive predictive value of 74% vs. 60%.[9] The technology was presented at European Society of Cardiology (ESC) by Dr. S. Seneviratne and at Radiological Society of North America (RSNA) and the American Heart Association (AHA). Using the technology for ED patients offers potential advantage over the HeartFlow process, because the turnaround time for the procedure is one to three hours. However, the early positive findings need to be validated with a more robust study.

Preclinical Data:

While few publications regarding the use of CT-FFR specifically address the cost of diagnostic work-up for obstructive disease, it is clear that the cost structure resulting from changes in diagnostic testing will also change. Deferral or avoidance of cardiac catheterization and nuclear stress testing will likely yield significant reductions in the cost of the diagnostic testing. In addition, because the results of the CT-FFR are available in the ED, CT-FFR has the potential to offer financial savings from reduced length of stay, while increasing patient satisfaction and reducing exposure to increased risk related to the emergency department environment.

Clinical Data to Date:

From 1/1/2009 to 3/31/2015 the investigative team introduced and operated a CCTA Chest Pain triage program for low to intermediate risk patients at Stony Brook University Hospital ED and non-emergency outpatient services, the only tertiary care hospital in Suffolk County, New York (NY). Concurrently, the investigators established a registry to monitor patient outcomes for all patients receiving CCTA at Stony Brook Medicine. The registry contained nearly 15,000 patient CCTA procedures. The major registry study established the effectiveness of CCTA as an imaging modality for evaluating ED chest pain in a cost efficient manner with a false negative rate less than 1% [5]. However, the registry reflects the poorer positive predictive values documented by other industry studies [6-8].

False positive workup results in the necessity of performing cardiac catheterization on patients at risk for obstructive disease based on assessment with current standard of care (combined screening with CCTA and stress MPI). Reduction in the rate of false positive testing would lead to reduction in risk from invasive procedures and radiation exposure to patients and reduced cost to the health care system.

Study Objectives:

The purpose of this study is to evaluate the incremental benefit of Fractional Flow Reserve derived from CCTA (FFR-CT) compared to invasive FFR as the gold standard for patients with obstructive disease (generally, >= 30% stenosis).

General Study Design:

This will be a prospective clinical trial designed to evaluate the incremental benefit of virtual FFR measured from CCTA, compared to invasive FFR and CCTA alone for the detection of flow-limiting coronary stenosis, as defined by invasive FFR <=0.8 and vessel diameter of >=2mm.

1,142 consecutive patients who present to North Shore University Hospital Emergency Department (ED) for CCTA due to chest pain or angina over a two year period and meeting the study inclusion criteria are eligible for the study (Figure 1). The investigators will employ CCTA-appropriateness criteria to ensure proper selection of patients, derived from the Appropriate Use Criteria for Cardiac Computed Tomography published in 2010 and jointly authored by multiple societies including American College of Cardiology Foundation (ACCF), Society of Cardiovascular Computed Tomography (SCCT), and American College of Radiology (ACR) [11]. FFR-CT measurements will be performed following CCTA scan acquisition on software developed by Toshiba America Medical Systems, Inc. All eligible patients will undergo 320-slice multi detector CCTA and CT-FFR measurements. The severity of the stenosis will be determined on site by level III CCTA readers.

Patients with borderline (50% - 70%) or positive CCTA (>70%) stenosis readings will undergo ICA with invasive FFR measurement in accordance with accepted guidelines and established practice standard. Those patients with invasively measured FFR<=0.8 and with vessel diameter of >= 2mm, or those who require revascularizations based on invasively estimated stenosis severity (for patients who are totally obstructed) will be considered to have flow-limiting obstructive CAD, while the rest will be considered to have non-flow limiting obstructive CAD (if also >50% stenosis on ICA). If stenosis severity turns out to be < 50% after ICA, these patients will have been shown to have non-obstructive CAD. (Figure 1). Patients with 30% to 49% obstructive stenosis by CCTA standards and with positive CT-FFR, will also undergo invasive FFR and follow the protocol for those with > 50% obstruction. Patients with 0 to 49% obstructive disease and negative CT-FFR will be referred to optimal follow up care only.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving informed consent.
2. Able to cooperate with the technician performing the procedure.
3. Patient must have Body Mass Index (BMI) <= 50.
4. Patients must have non-ST Elevation Myocardial Infarction (STEMI) Electrocardiogram (EKG) without acute changes.
5. Patients must present to North Shore University Hospital ED with Acute Chest Pain and require evaluation of coronary stenosis for the provisional diagnoses of acute chest pain or unstable angina or angina equivalent, and meet the criteria for CCTA by Heart Score Triage for the purpose of evaluation coronary stenosis for the provisional diagnoses of chest pain or angina or angina equivalent.

7.Patients must be able to take nitroglycerin and beta blockers. - 8.Patients must be 18 years of age or older.

Exclusion Criteria:

1. Patients must not have a history of coronary stenting or coronary artery bypass graft.
2. Patients must not have severe or end stage renal disease as diagnosed as estimated glomerular filtration rate (eGFR)<50.
3. Patients must not have a BMI>50.
4. Patient must not have any allergies to contrast.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Low to intermediate risk chest pain patients (as defined by the criteria above presenting to North Shore University Hospital, Northwell Health, Manhasset, NY for emergent assessement of chest pain symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 1142 (Estimated)
Dates: Start 2018-04-18 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of CT-FFR to Invasive FFR | Up to 2 years from the study initiation will be required to enroll all study patients and obtain invasive and noninvasive FFR.
  To evaluate sensitivity, specificity, positive and negative predictive value for CT-FFR, compared to invasive FFR.

SECONDARY OUTCOMES:
Return Visits | Up to 27 months will be required to collect 90 day follow up information on all study participants.
  To identify factors influencing return visits within 90 days for patient who had negative CCTA or Cardiac Catheterization findings.
Economic Impact | Up to 27 months will be requires to collect medical utilization after having administered CT-FFR
  To Compare the cost of care using CT-FFR by evaluating potentially avoidable workup with stress testing and invasive FFR.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Poon, MD, Principal Investigator — Northwell Health; Shahryar Saba, MD, Study Director — Northwell Health; Amar Shah, MD, Study Director — Northwell Health
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No
No Individual Participant Data (IPD) will be shared with other researchers. All study data will be deidentified to protect individual study participants identity.

REFERENCES:
- [Background] Min JK, Leipsic J, Pencina MJ, Berman DS, Koo BK, van Mieghem C, Erglis A, Lin FY, Dunning AM, Apruzzese P, Budoff MJ, Cole JH, Jaffer FA, Leon MB, Malpeso J, Mancini GB, Park SJ, Schwartz RS, Shaw LJ, Mauri L. Diagnostic accuracy of fractional flow reserve from anatomic CT angiography. JAMA. 2012 Sep 26;308(12):1237-45. doi: 10.1001/2012.jama.11274. PMID 22922562
- [Background] Norgaard BL, Leipsic J, Gaur S, Seneviratne S, Ko BS, Ito H, Jensen JM, Mauri L, De Bruyne B, Bezerra H, Osawa K, Marwan M, Naber C, Erglis A, Park SJ, Christiansen EH, Kaltoft A, Lassen JF, Botker HE, Achenbach S; NXT Trial Study Group. Diagnostic performance of noninvasive fractional flow reserve derived from coronary computed tomography angiography in suspected coronary artery disease: the NXT trial (Analysis of Coronary Blood Flow Using CT Angiography: Next Steps). J Am Coll Cardiol. 2014 Apr 1;63(12):1145-1155. doi: 10.1016/j.jacc.2013.11.043. Epub 2014 Jan 30. PMID 24486266
- [Background] Ko BS, Cameron JD, Meredith IT, Leung M, Antonis PR, Nasis A, Crossett M, Hope SA, Lehman SJ, Troupis J, DeFrance T, Seneviratne SK. Computed tomography stress myocardial perfusion imaging in patients considered for revascularization: a comparison with fractional flow reserve. Eur Heart J. 2012 Jan;33(1):67-77. doi: 10.1093/eurheartj/ehr268. Epub 2011 Aug 2. PMID 21810860
- [Background] Niska R, Bhuiya F, Xu J. National Hospital Ambulatory Medical Care Survey: 2007 emergency department summary. Natl Health Stat Report. 2010 Aug 6;(26):1-31. PMID 20726217
- [Background] Poon M, Cortegiano M, Abramowicz AJ, Hines M, Singer AJ, Henry MC, Viccellio P, Hellinger JC, Ferraro S, Poon A, Raff GL, Voros S, Farkouh ME, Noack P. Associations between routine coronary computed tomographic angiography and reduced unnecessary hospital admissions, length of stay, recidivism rates, and invasive coronary angiography in the emergency department triage of chest pain. J Am Coll Cardiol. 2013 Aug 6;62(6):543-52. doi: 10.1016/j.jacc.2013.04.040. Epub 2013 May 15. PMID 23684682
- [Background] Budoff MJ, Dowe D, Jollis JG, Gitter M, Sutherland J, Halamert E, Scherer M, Bellinger R, Martin A, Benton R, Delago A, Min JK. Diagnostic performance of 64-multidetector row coronary computed tomographic angiography for evaluation of coronary artery stenosis in individuals without known coronary artery disease: results from the prospective multicenter ACCURACY (Assessment by Coronary Computed Tomographic Angiography of Individuals Undergoing Invasive Coronary Angiography) trial. J Am Coll Cardiol. 2008 Nov 18;52(21):1724-32. doi: 10.1016/j.jacc.2008.07.031. PMID 19007693
- [Background] Meijboom WB, Meijs MF, Schuijf JD, Cramer MJ, Mollet NR, van Mieghem CA, Nieman K, van Werkhoven JM, Pundziute G, Weustink AC, de Vos AM, Pugliese F, Rensing B, Jukema JW, Bax JJ, Prokop M, Doevendans PA, Hunink MG, Krestin GP, de Feyter PJ. Diagnostic accuracy of 64-slice computed tomography coronary angiography: a prospective, multicenter, multivendor study. J Am Coll Cardiol. 2008 Dec 16;52(25):2135-44. doi: 10.1016/j.jacc.2008.08.058. PMID 19095130
- [Background] Ko BS, Cameron JD, Munnur RK, Wong DTL, Fujisawa Y, Sakaguchi T, Hirohata K, Hislop-Jambrich J, Fujimoto S, Takamura K, Crossett M, Leung M, Kuganesan A, Malaiapan Y, Nasis A, Troupis J, Meredith IT, Seneviratne SK. Noninvasive CT-Derived FFR Based on Structural and Fluid Analysis: A Comparison With Invasive FFR for Detection of Functionally Significant Stenosis. JACC Cardiovasc Imaging. 2017 Jun;10(6):663-673. doi: 10.1016/j.jcmg.2016.07.005. Epub 2016 Oct 19. PMID 27771399
- [Background] Miller JM, Rochitte CE, Dewey M, Arbab-Zadeh A, Niinuma H, Gottlieb I, Paul N, Clouse ME, Shapiro EP, Hoe J, Lardo AC, Bush DE, de Roos A, Cox C, Brinker J, Lima JA. Diagnostic performance of coronary angiography by 64-row CT. N Engl J Med. 2008 Nov 27;359(22):2324-36. doi: 10.1056/NEJMoa0806576. PMID 19038879
- [Background] Taylor AJ, Cerqueira M, Hodgson JM, Mark D, Min J, O'Gara P, Rubin GD; American College of Cardiology Foundation Appropriate Use Criteria Task Force; Society of Cardiovascular Computed Tomography; American College of Radiology; American Heart Association; American Society of Echocardiography; American Society of Nuclear Cardiology; North American Society for Cardiovascular Imaging; Society for Cardiovascular Angiography and Interventions; Society for Cardiovascular Magnetic Resonance; Kramer CM, Berman D, Brown A, Chaudhry FA, Cury RC, Desai MY, Einstein AJ, Gomes AS, Harrington R, Hoffmann U, Khare R, Lesser J, McGann C, Rosenberg A, Schwartz R, Shelton M, Smetana GW, Smith SC Jr. ACCF/SCCT/ACR/AHA/ASE/ASNC/NASCI/SCAI/SCMR 2010 appropriate use criteria for cardiac computed tomography. A report of the American College of Cardiology Foundation Appropriate Use Criteria Task Force, the Society of Cardiovascular Computed Tomography, the American College of Radiology, the American Heart Association, the American Society of Echocardiography, the American Society of Nuclear Cardiology, the North American Society for Cardiovascular Imaging, the Society for Cardiovascular Angiography and Interventions, and the Society for Cardiovascular Magnetic Resonance. J Am Coll Cardiol. 2010 Nov 23;56(22):1864-94. doi: 10.1016/j.jacc.2010.07.005. PMID 21087721
- [Result] Koo BK, Erglis A, Doh JH, Daniels DV, Jegere S, Kim HS, Dunning A, DeFrance T, Lansky A, Leipsic J, Min JK. Diagnosis of ischemia-causing coronary stenoses by noninvasive fractional flow reserve computed from coronary computed tomographic angiograms. Results from the prospective multicenter DISCOVER-FLOW (Diagnosis of Ischemia-Causing Stenoses Obtained Via Noninvasive Fractional Flow Reserve) study. J Am Coll Cardiol. 2011 Nov 1;58(19):1989-97. doi: 10.1016/j.jacc.2011.06.066. PMID 22032711